CLINICAL TRIAL: NCT01374672
Title: Observational - Methylation Status as Predictor of Response to Neoadjuvant Chemotherapy in Osteosarcoma
Brief Title: Biomarkers in Predicting Response to Chemotherapy in Samples From Young Patients With Osteosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AOST11B1; NCI-2011-02861 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-06-15; First posted 2011-06-16 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Localized Osteosarcoma; Metastatic Osteosarcoma; Osteoblastic Osteosarcoma; Recurrent Osteosarcoma
MeSH Terms: conditions — Osteosarcoma; Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative studies: DNA and RNA extracted from biopsy samples are analyzed for methylation changes and transcription changes by ligation-mediated PCR and mass-array genotyping.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research study is studying biomarkers in predicting response to chemotherapy in samples from young patients with osteosarcoma. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

DETAILED DESCRIPTION:
Study Subtype: Ancillary/Correlative Observational Study Model: Cohort Time Perspective: Retrospective Biospecimen Retention: Samples With DNA Biospecimen Description: Tissue Study Population Description: Children's Oncology Group Sampling Method: Non-Probability Sample

PRIMARY OBJECTIVES:

I. Determine whether methylation status predicts response to neoadjuvant chemotherapy in samples from children and young adults with osteosarcoma.

OUTLINE: Patients are stratified according to response to neoadjuvant chemotherapy (good vs poor).

DNA and RNA extracted from biopsy samples are analyzed for methylation changes and transcription changes by ligation-mediated PCR and mass-array genotyping.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with high-grade osteoblastic osteosarcoma
* Biopsy samples from patients who had good or poor response to neoadjuvant chemotherapy available
* All specimens should be from post-menarchal females or age-matched males with appendicular tumors
* Patients' clinical data including chemotherapy received, event-free survival, and overall survival available
* See Disease Characteristics

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosed with high-grade osteoblastic osteosarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Methylated status as predictor of response to neoadjuvant chemotherapy | Baseline
  Performed on a locus-by-locus basis using Poisson regression (for count data) and/or two-group t-tests, with correction (Satterwaithe's) for unequal within-group variances.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Rosenblum, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States